CLINICAL TRIAL: NCT00790231
Title: Effects of Thoracic Epidural Anesthesia on Lower Urinary Tract Function
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Patrick Yves Wüthrich/ Dr, Universitätsklinik für Anästhesiologie und Shcmerztherapie
Other Study IDs: KEK_105_08
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Urodynamics; Acute Urinary Retention
Keywords: urinary bladder; thoracic epidural analgesia; urodynamics; open kidney surgery with lumbotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- men: observation of the urinary function with and without thoracic epidural anesthesia
  Interventions: Device: urodynamic procedure
- women: observation of the urinary function with and without thoracic epidural anesthesia
  Interventions: Device: urodynamic procedure

INTERVENTIONS:
Device: urodynamic procedure — introduction of the urodynamic catheter into the bladder and assessment of the bladder function

SUMMARY:
Acute urinary retention is one of the most common complications after surgery and anesthesia. Overfilling the bladder can stretch and damage the detrusor muscle, leading to atony of the bladder. It can occur in patients of both sexes and all age groups and after all types of surgical procedures. Micturition depends on coordinated actions between the detrusor muscle and the external urethral sphincter. Motorneurons of both muscles are located in the sacral spinal cord and coordination between then occurs in the pontine tegmentum of the caudal brain stem. Motorneurons innervating the external urethral sphincter are located in the nucleus of Onuf, extending from the S1 to the S3 segment. The smooth detrusor muscle is inner-vated by parasympathetic fibers, which reside in the sacral intermediolateral cell group and are located in S2-4. Sympathetic fibers innervating the bladder and urethra play an important role in promoting conti-nence and are located in the intermediolateral cell group of the lumbar cord (L1-L4). Most afferent fibers from the bladder enter the sacral cord through the pelvic nerve at segments L4-S2 and the majority are thin myelinated or unmyelinated. Because peridural anesthesia can be performed at various levels of the spinal cord and with varying concentrations of local anesthetic, it is possible to block only a portion of the spinal cord (segmental blockade). So it seems logical that peridural analgesia from a Th 2-4 to Th 10-12 will have no influence on the micturition reflex. Studies on the urodynamic effects of various anaesthetic agents are rare. Under the influence of epidural analgesia, patients may not feel the urge to urinate, which may result in urinary retention and bladder over distension. Spinal and epidural opioid administrations influence the function of the lower urinary tract by direct spinal action on the sacral nociceptive neurons and autonomic fibres. It is therefore a common practice for bladder catheterisation in the presence of spinal or epidural anesthesia. The excessive use of a transurethral catheter is undoubtedly associated with significant morbidity such patient discomfort, urinary tract infections, catheter entrapment, bladder calculi formation, urethral trauma and stricture. The risk of infection with a single catheterization is 1-2% and can rise to 3 to 7 % a day. There has yet been no consensus for appropriate catheterisation strategy and urodynamic changes under thoracic epidural anesthesia are still unknown. We expect that a better knowledge on the bladder function under epidural analgesia could lead to a more restrictive use of perioperative transurethral catheters. Our hypothesis is that thoracic epidural analgesia does not influence lower urinary tract function in the male and female. Therefore transurethral catheterization is not mandatory for all patients with thoracic epidural analgesia. Differences in post void residual urine volume and urodynamic examinations before and during thoracic epidural analgesia will be analyzed in 16 men and 16 women undergoing open kidney surgery/lumbotomy who receive thoracic epidural anesthesia perioperatively.

DETAILED DESCRIPTION:
Acute urinary retention is one of the most common complications after surgery and anesthesia. It can occur in patients of both sexes and all age groups and after all types of surgical procedures. It is linked to several factors including increased intravenous fluids, postoperative pain and type of anesthesia. Micturition depends on coordinated actions between the detrusor muscle and the external urethral sphincter. Motorneurons of both muscles are located in the sacral spinal cord and coordination between them occurs in the pontine tegmentum of the caudal brain stem. Motorneurons innervating the external urethral sphincter are located in the nucleus of Onuf, extending from the S1 to the S3 segment. The detrusor smooth muscle is innervated by parasympathetic fibers, which reside in the sacral intermediolateral cell group and are located in S2-4. Sympathetic fibers innervating the bladder and urethra play an important role in promoting continence and are located in the intermediolateral cell group of the lumbar cord (L1-L4). Most afferent fibers from the bladder enter the sacral cord through the pelvic nerve at segments L4-S2 and the majority are thin myelinated or unmyelinated. nlike spinal anesthesia, which is an all or none block, epidural anesthesia has applications ranging from analgesia with minimal motor block to dense anesthesia (differential blockade). Because epidural anesthesia can be performed at various levels of the spinal cord, it is possible to block only a portion of the spinal cord (segmental blockade). Therefore it can be assumed that epidural analgesia within segments Th 4-6 to Th 10-12 has no or minimal influence on the micturition reflex. There are few studies on the urodynamic effects of various anaesthetic agents, focused on lumbar epidural anaesthesia. Under the influence of epidural analgesia, patients may not feel the urge to urinate, which can result in urinary retention and bladder overdistension. Overfilling of the bladder can stretch and damage the detrusor muscle. For example, the use of lumbar epidural analgesia for labor and delivery has frequently been implicated as a causative factor for postpartum urinary retention. This is supported by the fact that these patients demonstrate a difficulty voiding. Spinal and epidural opioid administration influence the function of the lower urinary tract by direct spinal action on the sacral nociceptive neurons and autonomic fibres. Long acting local anesthetics administrated intrathecally rapidly block the micturition reflex. Detrusor contraction is restored approximately 7-8 hours after spinal injection of bupivacaine. For this reason, bladder catheterisation is a common practice in patients with spinal or epidural anesthesia.The use of a transurethral catheter is associated with significant morbidity such as patient discomfort, urinary tract infections, urethral trauma and stricture. The risk of infection with a single catheterization is 1-2% and can rise by 3 to 7 % for every additional day with a indwelling catheter. Traumatic or prolonged catheterization may lead to urethritis and to urethral strictures. There has yet been no consensus for appropriate catheterisation strategy during regional anesthesia. We expect that a better knowledge on the bladder function under epidural analgesia could lead to a more restrictive use of perioperative transurethral catheters.Urodynamic changes under thoracic epidural anaesthesia are still unknown. The aim of this study is to compare lower urinary tract function before and during thoracic epidural analgesia within segments Th4-6 to Th 10-12 for postoperative pain treatment in patients undergoing lumbotomy for kidney surgery.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Open kidney surgery with lumbotomy
* Thoracic epidural analgesia

Exclusion Criteria:

* Significant renal dysfunction (creatinin >200mol/l)
* Contraindications to epidural anesthesia or refusal
* Preoperative residual urine volume > 100ml
* International Prostate Symptom Score (IPSS) > 7
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: open kidney surgery with lumbotomy, thoracic epidural analgesia
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Differences in postvoid residual urine volume before and during thoracic epidural analgesia | first measure preoperative, second measure on day 2 or 3 after surgeryx

SECONDARY OUTCOMES:
Bladder volume at first desire to void | first measure preoperative, second measure on day 2 or 3 after surgery
Bladder compliance | first measure preoperative, second measure on day 2 or 3 after surgery
Maximum detrusor pressure | first measure preoperative, second measure on day 2 or 3 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fiona C Burkhard, Prod, Study Chair — Dep. of Urology, Bern University Hospital; Patrick Y Wüthrich, MD, Principal Investigator — Dep. of Anesthsiology, Bern University Hospital
Locations (1):
- Department of Urology, Bern University Hospital, Bern, Switzerland